CLINICAL TRIAL: NCT06712719
Title: Effects of Dietary Phosphorus on Phosphorus and Calcium Whole-Body Balance and Kinetics in Moderate CKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: TBD2
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: CKD

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CKD patients group 1 (Experimental): assigned to Low P Diet (LP) then High P Diet (HP),
  Interventions: Other: LP then HP
- CKD patients group 2 (Experimental): assigned to HP, then LP.
  Interventions: Other: HP then LP

INTERVENTIONS:
Other: LP then HP — Cross-over order of LP then HP diet. Each cross-over phase will be 19 days and consist of a 7-day outpatient, controlled diet period, followed by a 5-day inpatient, controlled diet, balance, and kinetic study period, followed by a second 7-day outpatient, controlled diet period.
  Arms: CKD patients group 1
Other: HP then LP — Cross-over order of HP then LP diet. Each cross-over phase will be 19 days and consist of a 7-day outpatient, controlled diet period, followed by a 5-day inpatient, controlled diet, balance, and kinetic study period, followed by a second 7-day outpatient, controlled diet period.
  Arms: CKD patients group 2

SUMMARY:
The aim of the study is to look at the effects of dietary phosphorus on phosphorous and calcium whole-body balance and kinetics in moderate chronic kidney disease (CKD). N = 14 enrolled subjects will be randomly assigned to a cross-over order of (A) Low P Diet, High P Diet. Each cross-over phase will be 19 days and consist of a 7-day outpatient, controlled diet period, followed by a 5- day inpatient, controlled diet, balance, and kinetic study period, followed by a second 7-day outpatient, controlled diet period.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) affects approximately 37 million (1 in 7) U.S. adults, most of whom experience mineral and bone disorders (CKD-MBD) that increase risk for cardiovascular events, bone fractures, and death. Dietary and pharmaceutical treatments for CKD-MBD have diverse effects on serum calcium and phosphorus levels, but their effects on the underlying physiological processes of calcium and phosphorus balance are largely unknown. This study aims to determine the effects of a low versus high phosphorus bioaccessibility diet on whole-body calcium and phosphorus balance and kinetics, including measures such as estimated intestinal absorption. This study will be a randomized two-phase cross-over design trial that will include a controlled study diet, a phosphorus isotope as a tracer for kinetic modeling, stool and urine collections, and blood draws. After screening, eligible participants who choose to enroll in the study will be asked to participate in two cross-over sessions, each of approximately 3 weeks (19 days) duration during which time all food will be provided according to the randomized diet intervention assignment. After the first week on the study diet, participants will be asked to stay at the clinical research center when they will be given oral and intravenous doses of phosphorus isotope. Serial blood draws and complete urine and fecal collections will be made for 5 days, then the final week will only include blood draws. Between cross-over sessions, there will be a washout period of 1-3 weeks. Participants will then switch diets and repeat the same study process as the first session. Calcium and phosphorus whole-body balance, intestinal absorption, renal excretion, and movement to and from bone will be determined for both minerals. This project will provide foundational knowledge of calcium and phosphorus physiology in CKD that will support progress towards preventing morbidity and mortality associated with CKD-MBD.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, ages 30-75 years old, any race or ethnicity
* Moderate CKD, defined by KDIGO as eGFR category 3b (30-44 mL/min) or 4 (16-29 mL/min) with albuminuria categories A1-A3
* Serum intact parathyroid hormone above assay normal limit
* Female subjects must be postmenopausal (>12 months since last menstrual period), surgically sterile, or confirmed not pregnant by pregnancy test
* Must be on stable doses of medications (except those noted in exclusion criteria) for at least 4 weeks prior to the study
* Willing to discontinue supplements (e.g., vitamin D, calcium, multivitamin/minerals, or others) upon enrollment until completion of the study
* Adequate vitamin D status defined as serum 25D > 20 ng/mL based on National Academy of Medicine (then Institute of Medicine) criteria.

Exclusion Criteria:

* Plans to initiate dialysis within 6 months
* Hypercalcemia defined as corrected serum calcium >9.8 mg/dL within past 3 months
* Hyperkalemia defined as serum potassium >5.5 mg/dL within past 3 months
* Hyperphosphatemia defined as serum phosphate >5.5 mg/dL within past 3 months
* Intestinal disease that alters absorption or normal intestinal function including celiac disease, small bowel resection, bariatric surgery, or chronic diarrhea/malabsorption
* Serious, uncontrolled underlying systemic disease including diabetes, lupus, hypertension in the opinion of their physician
* Pregnant or breastfeeding
* Prescribed and taken a phosphate binder medication, calcitriol, vitamin D analogs, calcimimetics, PTH analogues, and other medications that may alter Ca and P metabolism within past 4 weeks
* Non-English speaking

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-05-28 (Estimated); Study Completion 2027-05-28 (Estimated)

PRIMARY OUTCOMES:
Phosphorus Balance | 5 days
  Determined by analysis of phosphorus content in complete 24-hour urine and stool collections, subtracted from the diet phosphorus content consumed
Calcium Balance | 5 days
  Determined by analysis of calcium content in complete 24-hour urine and stool collections, subtracted from the diet calcium content consumed

SECONDARY OUTCOMES:
Fractional phosphorus absorption | 12 days
  Determined by kinetic modeling of serum, urine, and stool P-33 isotope after oral and IV isotope administrations
Bone phosphorus balance | 12 days
  Determined by kinetic modeling of serum, urine, and stool P-33 isotope after oral and IV isotope administrations
Bone calcium balance | 5 days and 12 days
  Determined from the natural stable isotope ratio of 44-Ca to 42-Ca in serum and urine
Urine phosphorus | 1 week
  Determined from the 24-hour urine collections over 1 week (daily average)
Urine calcium | 1 week
  Determined from the 24-hour urine collections over 1 week (daily average)
Net phosphorus absorption | 1 week
  Determined by analysis of phosphorus content in complete stool collections, subtracted from the diet phosphorus content consumed, divided by the diet phosphorus consumed.
Net calcium absorption | 1 week
  Determined by analysis of calcium content in complete stool collections, subtracted from the diet calcium content consumed, divided by the diet phosphorus consumed
Creatinine clearance | 2hours, day 8
  Creatinine clearance will be determined from the 2-hour fasting urine and a mid-point blood sample collected on Day 8.
Serum Fibroblast growth factor-23 | Day1, Day8
  Measured in a fasting blood collection on Day 1 and Day 8.
Serum Parathyroid hormone | Day1, Day8
  Measured in a fasting blood collection on Day 1 and Day 8.
Serum 1,25-dihydroxyvitamin D | Day1, Day8
  Measured in a fasting blood collection on Day 1 and Day 8.
Serum phosphate | Day1, Day8
  Measured in a fasting blood collection on Day 1 and Day 8.
Serum calcium | Day1, Day8
  Measured in a fasting blood collection on Day 1 and Day 8.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Hill Gallant, PhD, Principal Investigator — University of Minnesota